CLINICAL TRIAL: NCT02212600
Title: The DECIPHER Study: Determinants of Function and Clinically Important Outcomes in Proximal Humerus Fractures in the Elder Population: A National Cohort
Brief Title: Determinants of Function and Clinically Important Outcomes in Proximal Humerus Fractures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Emil Schemitsch, MD, FRCSC, London Health Sciences Centre
Other Study IDs: DECIPHER
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Humeral Fractures, Proximal
MeSH Terms: conditions — Shoulder Fractures | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Population: We will include male and female patients who are over 50 years of age and who have an acute, displaced or undisplaced proximal humerus fracture caused by low energy trauma
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — observational cohort of proximal humerus fractures

SUMMARY:
The proposed project will be a multi-centre, prospective observational study to determine the prognosis and determinants of functional outcomes of patients with proximal humerus fractures. Approximately 10 centres will participate in this observational cohort, each enrolling at least 50 patients over the course of 2 years.

ELIGIBILITY:
Inclusion Criteria:

males and females age 50 years or older (no uper age limit) presenting with an acute displaced or undisplaced proximal humerus fracture

Exclusion Criteria:

pathologic fractures patients likely to be lost before completing follow-up patients who do not provide consent patients who do not speak English and who do not have a translator that will be available during consent discussion and at each follow-up.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will include male and female patients who are over 50 years of age and who have an acute, displaced or undisplaced proximal humerus fracture caused by low energy trauma and who provide written informed consent.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-09-10 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder, and Hand (DASH) | 2 years
  The DASH is a 30-item, self-report questionnaire designed to measure physical function and symptoms in people with musculoskeletal disorders of the upper limb.

SECONDARY OUTCOMES:
Rate of complications | 2 years
  Clinical outcomes will include range of motion measurements, standardized radiographic evaluation, assessment of complications, rate of re-operation, infections, osteonecrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Emil Schemitsch, MD, FRCSC, Principal Investigator — London Health Scieneces Centre and St. Michael's Hospital
Locations (2):
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario